CLINICAL TRIAL: NCT01853176
Title: Is Liposomal Injection Bupivacaine (Exparel) Superior to Standard Bupivacaine for Abdominoplasty? A Randomized Controlled Trial
Brief Title: Exparel vs. Standard Bupivicaine for Abdominoplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: required documentation too onerous
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Albert Losken, MD, Professor, Division of Plastic Surgery, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00064693
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Pain, Postoperative
Keywords: Pain, Postoperative; Analgesia; Anesthesia, local; Abdominoplasty
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposomal injection bupivicaine (Exparel) (Experimental): Patients will have the maximum approved dose of Exparel, 266 mg, diluted in 20 mL normal saline, infiltrated into the rectus fascia and subcutaneous tissues at the time of abdominoplasty.
  Interventions: Drug: Liposomal Injection Bupivacaine (Exparel)
- Standard bupivicaine (Active Comparator): Patients will receive the maximum safe allowance of 0.25% bupivacaine, or 1.5 mg/kg (eg. 150 mg or 60 mL for a 100 kg patient) infiltrated into the rectus fascia and subcutaneous tissues at the time of abdominoplasty.
  Interventions: Drug: Standard bupivicaine

INTERVENTIONS:
Drug: Liposomal Injection Bupivacaine (Exparel)
  Other Names: Exparel; bupivicaine liposome injectable suspension
  Arms: Liposomal injection bupivicaine (Exparel)
Drug: Standard bupivicaine
  Other Names: bupivicaine; Marcaine
  Arms: Standard bupivicaine

SUMMARY:
Background & study question:

Strategies for post-operative pain control that make use of various different types of medicines are advantageous both for patient comfort and for minimizing the use of opioid pain medicines and their associated side effects, which include drowsiness, nausea, and vomiting. A key element of these strategies is wound injection with local anesthetic (numbing medicine) at the time of surgery. Local numbing procedures are used routinely in patients undergoing abdominoplasty (tummy tuck), most often with lidocaine or bupivacaine, which can last several hours. Multiple studies have shown that locally injected pain medicines achieve better pain control, less opioid use, and faster return to normal activities, such that the use of one of these local anesthetic medicines is the current standard of care.

Exparel is an extended-release formulation of bupivacaine that can produce local pain relief for up to 72 hours. Studies have shown it to provide better post-operative pain control and decreased use of opioid medications when compared to patients who did not receive any local numbing agents. Exparel has been used successfully in a variety of surgical settings, including open colon surgery, laparoscopic gall bladder removal, abdominoplasty, and breast augmentation. Its effectiveness has by and large been established in comparison to no local anesthetic. In this study, we seek to investigate the benefit of Exparel compared to standard bupivacaine infiltration in patients undergoing abdominoplasty.

Study design:

Patients scheduled for abdominoplasty with the lead investigator will be offered inclusion in this study. Consenting patients will be randomly assigned to standard bupivacaine or Exparel by coin toss after their clinic visit. On the day of surgery, the only difference between patients assigned to one arm or the other is the local anesthetic used. The surgery itself and plan for general anesthesia will be similar. Both groups will have the same pain medicines available after surgery.

Patients will be given a form on which to record twice-daily pain ratings and opioid narcotic needs for 3 days after surgery. For patients admitted after surgery, oral and IV narcotic use will be collected from their inpatient medical record.

The primary outcome of interest is daily and cumulative pain scores through 3 days. A secondary endpoint is daily and total opioid use over 3 days. Additional measures include the time to first post-operative use of opioid medication and incidence of any adverse side effects.

ELIGIBILITY:
Inclusion Criteria:

* adult men and women
* scheduled for abdominoplasty

Exclusion Criteria:

* pregnant women
* patients with allergy to amide-type local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Losken, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory Aesthetic Center at Paces, Atlanta, Georgia

REFERENCES:
- [Background] Gorfine SR, Onel E, Patou G, Krivokapic ZV. Bupivacaine extended-release liposome injection for prolonged postsurgical analgesia in patients undergoing hemorrhoidectomy: a multicenter, randomized, double-blind, placebo-controlled trial. Dis Colon Rectum. 2011 Dec;54(12):1552-9. doi: 10.1097/DCR.0b013e318232d4c1. PMID 22067185
- [Background] Haas E, Onel E, Miller H, Ragupathi M, White PF. A double-blind, randomized, active-controlled study for post-hemorrhoidectomy pain management with liposome bupivacaine, a novel local analgesic formulation. Am Surg. 2012 May;78(5):574-81. doi: 10.1177/000313481207800540. PMID 22546131
- [Background] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785
- [Background] Chavez-Abraham V, Barr JS, Zwiebel PC. The efficacy of a lidocaine-infused pain pump for postoperative analgesia following elective augmentation mammaplasty or abdominoplasty. Aesthetic Plast Surg. 2011 Aug;35(4):463-9. doi: 10.1007/s00266-010-9633-4. Epub 2010 Dec 7. PMID 21136251
- [Background] Feng LJ. Painless abdominoplasty: the efficacy of combined intercostal and pararectus blocks in reducing postoperative pain and recovery time. Plast Reconstr Surg. 2010 Nov;126(5):1723-1732. doi: 10.1097/PRS.0b013e3181ef8fe5. PMID 21042130

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at Emory University Hospital - Midtown between October 2013 through November 2013.
Groups:
- Liposomal Injection Bupivicaine (Exparel): Patients will have the maximum approved dose of Exparel, 266 mg, diluted in 20 mL normal saline, infiltrated into the rectus fascia and subcutaneous tissues at the time of abdominoplasty.
  Liposomal Injection Bupivacaine (Exparel)
- Standard Bupivicaine: Patients will receive the maximum safe allowance of 0.25% bupivacaine, or 1.5 mg/kg (eg. 150 mg or 60 mL for a 100 kg patient) infiltrated into the rectus fascia and subcutaneous tissues at the time of abdominoplasty.
  Standard bupivicaine
Period: Overall Study
Arm/Group | Liposomal Injection Bupivicaine (Exparel) | Standard Bupivicaine
Started | 4 | 0
Completed | 0 | 0
Not Completed | 4 | 0
Not completed — Study terminated | 4 | 0

BASELINE CHARACTERISTICS:
Population: Did not meet target accrual before study terminated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Injection Bupivicaine (Exparel) | Standard Bupivicaine | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 4 |  | 4
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 4 |  | 4
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Pain Score, Visual Analogue Pain Scores
Description: Continuous Visual Analogue Scale 0 - 10 (0=no pain, 10=worst imaginable pain. Patients will complete a log of pain levels experienced each morning and evening for 3 days. Score is 0-10 on a visual analog scale.
Time Frame: 3 days
Arm/Group | Liposomal Injection Bupivicaine (Exparel) | Standard Bupivicaine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Liposomal Injection Bupivicaine (Exparel) | Standard Bupivicaine
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 0/0

LIMITATIONS AND CAVEATS:
Trial terminated prior to any meaningful patient accrual so no analysis performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes